CLINICAL TRIAL: NCT03408002
Title: PREPARE: Valutazione di un Intervento Psicologico Pre-operatorio in Pazienti Che Saranno Sottoposti a Chirurgia Del Pancreas
Brief Title: PREPARE - PREoPerative Anxiety REduction
Acronym: PREPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: University of Pisa (Other); Universita di Verona (Other)
Responsible Party: Principal Investigator, Lidia Del Piccolo, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Prog. 1288CESC
Record Dates: First submitted 2017-07-20; First posted 2018-01-23 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Anxiety Disorder; Surgery
Keywords: preoperative anxiety; self-efficacy; psychophysiology; psychotherapy; pancreatic surgery
MeSH Terms: conditions — Anxiety Disorders | interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): no intervention
- Psychological intervention (Experimental): Psychological intervention using the "Four elements" technique elaborated by Shapiro and reported in M. Luber (2009) during a psychological consultation conducted the day before surgery.
  Interventions: Behavioral: Psychological intervention

INTERVENTIONS:
Behavioral: Psychological intervention — The intervention aims to increase self-efficacy perception in managing pre-operative anxiety. The intervention is based on one single psychological consultation adopting the "Four elements" technique elaborated by Shapiro
  Arms: Psychological intervention

SUMMARY:
The study aims to verify if a short individual psychological intervention might increase perceived self-efficacy in managing preoperative anxiety in patients who will undergo pancreatic surgery. It is a randomized clinical trial where half of participants will attend a psychological intervention based on "the four elements protocol" by Elan Shapiro the day before surgery, while the other half will follow usual care.

DETAILED DESCRIPTION:
Patients who have to undergo surgery experience multiple sources of stress. A recent narrative review carried out on 115 studies by Powell et al. (2016) reported different and inconsistent findings on the relation between psychological interventions and surgery outcomes, due to the heterogeneity of these interventions, mainly based on information giving and patient education, and the very different samples of patients considered. Some evidences showed that pre-operative psychological interventions may contribute to reduce post-operative pain, duration of hospital stay (mean difference of 0.52 days) and negative affect. No studies were conducted with patients who had to undergo pancreatic surgery nor specific psychological interventions were devoted to increase self-efficacy in managing anxiety.

The aim of the present study is to verify if a short individual psychological intervention devoted to improve patient's ability to manage anxiety could increase his/her confidence to cope with pancreatic surgery, either in terms of perceived self-efficacy (main outcome) or less state anxiety reported on STAI-Y1 scale. Post-surgery outcomes are also collected: pain reported during the days following surgical intervention, length of hospital stay and number and type of clinical complications.

The study will involve 400 patients randomly divided in two arms and it is organized in four phases: T0,T1,T2,T3.

T0: Once obtained the informed consent, demographic information will be collected using a structured questionnaire. Clinical variables will be collected by self-administered tools, for which patients can ask support, if needed.

T1: The day before surgery, all patients will indicate their perceived self-efficacy in managing anxiety and will fulfil specific anxiety scales.

T2: after randomization, patients in the experimental group will participate to the psychological intervention, whereas the control group will follow usual care.

T3: After surgery pain, length of hospital stay and the number of post-operative complications within 30 days will be evaluated as secondary outcomes on all patients.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years old
* cognitively able to give personal consent to participate to the study
* to be scheduled to have general anaesthesia for pancreatic surgery

Exclusion Criteria:

* age under 18 years and over 80 years
* cognitively unable to give personal consent to participate to the study
* postponement of surgical operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change of Perceived self-efficacy, comparing the score on analogue scale (range 1-10) before (baseline) and after the psychological intervention in the experimental group. | Perceived self-efficacy will be measured before (baseline) and immediately after the psychological intervention (up to 1 hour) in the experimental group, whereas in the control group it will be measured only once (baseline).
  To measure perceived self-efficacy, patients respond to the following question: "We kindly ask you to indicate on a scale from 1 to 10 how much you perceive to be able to manage anxiety before the surgery".

SECONDARY OUTCOMES:
Post-operative pain measured by the Brief Pain Inventory | 3rd day after surgery
  It is a brief questionnaire composed which evaluates the intensity of perceived pain during the last 24 hours. The patient indicates on a human figure where is located the pain and its intensity on an analogue scale (range 1-10), then the patient responds to seven questions asking how this pain interferes with general activities, work, mood, ability to walk, quality of slumber and social relationships.
Number of perioperative complications | 30 days
  Description of the number and type of post-operative complications
Number of days of hospitalization | From date of hospital admission until the date of discharge or date of death from any cause, whichever came first, assessed up to 6 months.
  Exact number of hospitalization days for each patient
VAS-P Visual Analogue Scale of Pain. | from the 3rd day until 5th day after surgery
  VAS-P is a visual analogue scale where number 0 represents "absence of pain" and number 10 indicates "the worse pain ever tried". To measure perceived postoperative pain, patients respond to the following question: "We kindly ask you to indicate on a scale from 0 to 10 the intensity of your pain".The scale has no standardized scores or cut-off. Each patient applies his or her own "yardstick" in answering questions. Lower values are considered a better outcome.

OTHER OUTCOMES:
Preoperative Anxiety comparing the score before (baseline) and after the psychological intervention in the experimental group and only at baseline in the control group. | Preoperative Anxiety will be measured before (baseline) and immediately after the psychological intervention (up to 1 hour) in the experimental group, whereas in the control group it will be measured only once (baseline).
  Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a Likert (scoring from 1="not at all" to 5="completely agree") 6 item scale
Change of state anxiety, comparing the score before (baseline) and after the psychological intervention in the experimental group and only at baseline in the control group. | State anxiety will be measured before (baseline) and immediately after the psychological intervention (up to 1 hour) in the experimental group, whereas in the control group it will be measured only once (baseline).
  State-Trait Anxiety Inventory (STAI-Y1)
WAI-T, Therapist version of Working Alliance Inventory (Only experimental group) | Immediately after the conclusion of the psychological intervention (up to 1 hour)
  WAI-T is a 36-item Likert scale on 7 points. There is no cut-off. Higher values indicate a better outcome.
WAI-C, Client version of Working Alliance Inventory (Only experimental group) | Immediately after the conclusion of the psychological intervention (up to 1 hour)
  WAI-C is a 36-item Likert scale on 7 points.There is no cut-off. Higher values indicate a better outcome.
Electrodermal activity (Only experimental group patients without jaundice, feverish states, pancreatic pain with analgesic therapy, recent neoadjuvant therapy, psychotropic therapy or cardio-vascular problems will be included) | Collection during psychological intervention (which lasts on average one hour), after collecting 4 minutes of baseline.
  Skin Conductance Level (SCL) measured in microsiemens (μS), using the Biopac MP150 system, which is connected to a Windows 7 operated computer running Acknowledge 4.1 data acquisition program and Observer XT 10.0 (Noldus).
Heart Rate Variability (HRV) (Only experimental group patients without jaundice, feverish states, pancreatic pain with analgesic therapy, recent neoadjuvant therapy, psychotropic therapy or cardio-vascular problems will be included) | Collection during psychological intervention (which lasts on average one hour), after collecting 4 minutes of baseline.
  Beat-to-beat variation of heart rate over time. ECG signals will be recorded by means of ECG100C Electrocardiogram Amplifier from BIOPAC MP150 system, with a sampling rate of 500 Hz. BIOPAC is connected to a Windows 7 operated computer running Acknowledge 4.1 data acquisition program and Observer XT 10.0 (Noldus).

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Del Piccolo, Principal Investigator — Azienda Ospedaliera Universitaria Integrata
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, Italy

REFERENCES:
- [Derived] Marinelli V, Danzi OP, Mazzi MA, Secchettin E, Tuveri M, Bonamini D, Rimondini M, Salvia R, Bassi C, Del Piccolo L. PREPARE: PreoPerative Anxiety REduction. One-Year Feasibility RCT on a Brief Psychological Intervention for Pancreatic Cancer Patients Prior to Major Surgery. Front Psychol. 2020 Mar 5;11:362. doi: 10.3389/fpsyg.2020.00362. eCollection 2020. PMID 32194490